CLINICAL TRIAL: NCT00634361
Title: Ethyl-EPA Treatment of Prodromal Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA01.03.0011; NCT00237835 (obsolete NCT alias)
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia Prodrome
MeSH Terms: interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: ethyl-eicosapentaenoic acid

INTERVENTIONS:
Drug: ethyl-eicosapentaenoic acid — 2 mg per day
  Other Names: ethyl-EPA, an omega-3 fatty acid

SUMMARY:
This is an open-label trial of an omega-3 fatty acid for symptoms of the schizophrenia prodrome.

ELIGIBILITY:
Inclusion Criteria:

* meets criteria for schizophrenia prodrome

Exclusion Criteria:

* any lifetime antipsychotic treatment

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2001-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
conversion to psychosis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Yale University